CLINICAL TRIAL: NCT06459492
Title: Effect of Puzzle Game Strategy on Cognitive Functioning and Psychological Well-being Among Older Adults
Brief Title: Puzzle Game Strategy on Older Adults
Acronym: PUZZLEOLDER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 13620
Record Dates: First submitted 2024-05-19; First posted 2024-06-14 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-05

CONDITIONS: Old Age; Debility
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- puzzle game strategy study group (Experimental): Older adults who participate in puzzle game strategies
  Interventions: Behavioral: puzzle game strategies
- older adult control group (No Intervention): Older adults who not participate in puzzle game strategies

INTERVENTIONS:
Behavioral: puzzle game strategies — One innovative approach uses puzzle game strategies, including crosswords, Sudoku, and other brain-teasing activities. These strategies have been shown to help maintain attention, improve memory, and keep older adults' thoughts clear and sharp. Additionally, engaging in these activities can provide psychological benefits by offering a sense of achievement, reducing stress, and fostering social interactions.
  Given puzzle games' potential to enhance cognitive and psychological health, exploring their effectiveness as a non-pharmacological intervention for community-dwelling older adults is essential. This research aims to fill the gap by empirically investigating the impact of puzzle game strategies on cognitive functioning and psychological well-being in this demographic.
  Arms: puzzle game strategy study group

SUMMARY:
One innovative approach uses puzzle game strategies, including crosswords, Sudoku, and other brain-teasing activities. These strategies have been shown to help maintain attention, improve memory, and keep older adults' thoughts clear and sharp. Additionally, engaging in these activities can provide psychological benefits by offering a sense of achievement, reducing stress, and fostering social interactions.

DETAILED DESCRIPTION:
Cognitive abilities naturally decline as people age, one factor leading to deteriorating psychological health among older adults. Therefore, it is crucial to develop interventions to enhance this population's cognitive abilities and psychological well-being through non-pharmacological complementary treatments. Such interventions should focus on improving these symptoms while replacing traditional therapies.

One innovative approach uses puzzle game strategies, including crosswords, Sudoku, and other brain-teasing activities. These strategies have been shown to help maintain attention, improve memory, and keep older adults' thoughts clear and sharp. Additionally, engaging in these activities can provide psychological benefits by offering a sense of achievement, reducing stress, and fostering social interactions.

Given puzzle games' potential to enhance cognitive and psychological health, exploring their effectiveness as a non-pharmacological intervention for community-dwelling older adults is essential. This research aims to fill the gap by empirically investigating the impact of puzzle game strategies on cognitive functioning and psychological well-being in this demographic.

ELIGIBILITY:
Inclusion Criteria:

* Aged 60 years and above.
* Able to communicate effectively.
* Have mild or moderate cognitive impairment,

Exclusion Criteria:

* Have rheumatoid arthritis.
* Hand tremors that could limit their ability to use puzzles.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Older adults who participate in puzzle game strategies and cognitive functioning by Mental Health Scale (MHS) | three months
  Older adults who participate in puzzle game strategies will exhibit lower cognitive difficulties by MHS (scores ranging from 0 to 10, with a higher score indicating lower cognitive difficulties) than those who do not enter intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria university, Alexandria, Alexandria Governorate, Egypt